CLINICAL TRIAL: NCT01885221
Title: A Multi-Media Approach to Partner Support in Smokeless Tobacco Cessation
Brief Title: A Multi-Media Approach to Partner Support in Smokeless Tobacco Cessation (UCare-ChewFree)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA033422
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Tobacco Use Cessation
Keywords: smokeless tobacco cessation; social support; partner support
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multimedia Support Intervention (Experimental): (a) access to a website providing the content of our supporter guidebook, supplemented with interactive components, video elements, and a supporters' forum, and (b) a mailed copy of our supporter guidebook
  Interventions: Behavioral: Multimedia Support Intervention
- Delayed Treatment Control (No Intervention): Access to the Multimedia Intervention after participant completes the final follow-up assessment

INTERVENTIONS:
Behavioral: Multimedia Support Intervention
  Arms: Multimedia Support Intervention

SUMMARY:
In an earlier study, the investigators developed a guidebook that taught women supportive behaviors to help their husbands/partners quit smokeless tobacco. This study will create a website using the information in the guidebook, along with interactive features, videos, and forums. The investigators will then conduct a randomized trial comparing an intervention group (receiving website access and the printed guidebook) with a delayed treatment control condition, to learn if the support intervention can effectively teach women supportive behaviors and thereby increase their partners' smokeless tobacco cessation rates.

ELIGIBILITY:
Inclusion Criteria:

* being the wife or female domestic partner (living together) of a male who is a current user of ST products (snuff or chewing tobacco)
* interested in having him quit ST use
* willing to provide a phone number, mailing address, and e-mail address
* provides informed consent
* the woman and the chewer are both U.S. or Canadian residents age 18 or older
* the woman and the chewer are both able to read English
* the woman and the chewer are both able to access a computer

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
smokeless tobacco cessation | 7.5-month follow-up
  the male ST user's 6-month cessation as reported by the female partner

SECONDARY OUTCOMES:
tobacco quit attempts | 7.5 month follow-up
  the male smokeless tobacco user's quit attempts, as reported by the female partner
supportive behaviors | 7.5 month follow-up
  change in the female partner's supportive behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Laura E Akers, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

REFERENCES:
- [Derived] Akers L, Andrews JA, Lichtenstein E, Severson HH, Gordon JS. Effect of a Responsiveness-Based Support Intervention on Smokeless Tobacco Cessation: The UCare-ChewFree Randomized Clinical Trial. Nicotine Tob Res. 2020 Mar 16;22(3):381-389. doi: 10.1093/ntr/ntz074. PMID 31070741
- [Derived] Akers L, Andrews JA, Gordon JS. A Multimedia Support Skills Intervention for Female Partners of Male Smokeless Tobacco Users: Use and Perceived Acceptability. JMIR Form Res. 2018 Jan-Jun;2(1):e10. doi: 10.2196/formative.9948. PMID 30556053